CLINICAL TRIAL: NCT05606003
Title: Using a Community-level Just-in-Time Adaptive Intervention to Address COVID-19 Testing Disparities: A Population-based Study
Brief Title: Using a Community-level Just-in-Time Adaptive Intervention to Address COVID-19 Testing Disparities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Maria E Fernandez, Lorne Bain Distinguished Professorship in Public Health and Director, Center for Health Promotion and Prevention Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-SPH-20-1372 Main Study; 3UL1TR003167 (NIH)
Record Dates: First submitted 2022-09-19; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: COVID-19 testing; decision making; testing behaviors; vulnerable populations
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-level Multi-Component Intervention (MLI) (Experimental): Individuals receive COVID-19 CHW-delivered education and navigation, 2-1-1 helpline referrals, and social marketing messaging.
  Interventions: Behavioral: Multi-Level Multi-Component Intervention (MLI)
- Community Just-in-Time-Adaptive Intervention (JITAI) (Experimental): Individuals receive MLI intervention components that are informed by real-time data and community stakeholder feedback.
  Interventions: Behavioral: Community Just-In-Time Adaptive Intervention (Community JITAI)
- Comparison Condition (No Intervention): Individuals receive standard exposure to ongoing city and county COVID-19 communication and testing.

INTERVENTIONS:
Behavioral: Multi-Level Multi-Component Intervention (MLI) — The strategic components of our multi-level, multi-component intervention (MLI) include: 1. Building testing access for vulnerable populations, 2) Community Health Worker (CHW)-delivered navigation to SARSCoV- 2 testing and access and reinforce risk mitigation recommendations, 3) 2-1-1 helpline-referrals and navigation to FDA approved SARSCoV- 2 testing (and self sampling once approved) and risk mitigation education, and 4) social marketing and small media campaign to provide geo-targeted messages promoting testing and COVID risk mitigation behaviors. We selected these components because of their evidence base, their current use by partners in response to COVID 19, and confidence that they can be adapted through a community engaged process as described.
  Arms: Multi-level Multi-Component Intervention (MLI)
Behavioral: Community Just-In-Time Adaptive Intervention (Community JITAI) — This intervention includes the same MLI components described above, with an added JITAI approach. Community and stakeholder partners will use real-time data related to testing and other relevant information generated by the Epidemiologic Surveillance and Analysis team (ESA) in Aim 1, as well as other information based on their community and stakeholder experience and tacit knowledge about factors influencing testing determinants, to adapt intervention activities as needed to optimize access to testing.
  Arms: Community Just-in-Time-Adaptive Intervention (JITAI)

SUMMARY:
In collaboration with community partners, this study will identify disparities and dynamics of COVID-19 testing and infections in three Texas regions; and implement a multilevel intervention that increases access to testing and referrals to follow-up care among vulnerable populations. Using a three-arm group-randomized controlled trial, this study will assess the impact of multi-level interventions influencing motivation and access to testing.

The outcomes of this study are measured at the population level and no individual data will be gathered. Analyses of de-identified PHI data from local and regional health departments on COVID testing and infection rates will be used to assess intervention outcomes.

DETAILED DESCRIPTION:
In the U.S. vulnerable populations experience significant disparities in terms of both COVID-19 infection and mortality rates, especially in Texas, where Hispanic, African Americans, and other groups have experienced substantial disparities in both incidence and mortality. Building on the partnerships and resources of the Center for Clinical and Translational Science (CCTS), the goal of the proposed project is to identify dynamic COVID-19 disease hotspots and testing deserts in racially diverse regions of South Texas, Houston/Harris County, Texas, and Northeast Texas to inform the rapid adaptation and deployment of multilevel level just-in-time adaptive intervention strategies to reduce testing disparities among vulnerable populations.

A group-randomized controlled trial (RCT) will be conducted to evaluate the reach, effectiveness, and implementation of a community-level Just-In-Time-Adaptive-Intervention (JITAI) to increase COVID-19 testing in identified high-risk priority neighborhoods. To conduct the RCT, 120 priority census blocks groups will be identified and randomized to each condition using a community risk index score that balances distribution in the three study arms with respect to important characteristics including population density, demographics, and baseline testing rates.

In Intervention Condition 1 - Multi-Level Multi-Component Intervention (MLI), individuals will receive a multilevel, multi-component intervention comprising of 1) Building testing access for vulnerable populations, 2) Community Health Worker (CHW)-delivered navigation to COVID-19 testing and access and reinforcing risk mitigation recommendations; 3) 2-1-1 helpline-referrals and navigation to testing and 4) social marketing and small media campaign to provide geo-targeted messages promoting testing and COVID-19 risk mitigation behaviors. In Intervention Condition 2 - Community JITAI individuals will receive the same MLI intervention components but with an added JITAI approach informed by real-time data related to testing and other relevant information based on community and stakeholder experience and tacit knowledge about factors influencing testing determinants. The Comparison Condition will receive standard exposure to ongoing city and county communication and access to testing.

ELIGIBILITY:
Inclusion Criteria:

* residing in identified COVID-19 hotspots and testing deserts within study regions
* aged 18 years or older

Exclusion Criteria:

* aged under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Testing Uptake | Baseline through study completion (26 months)
  Examine the short and long-term change in testing proportion from baseline in the CBGs adjusted for testing capacity (testing proportion in the county during the same time period)

SECONDARY OUTCOMES:
Disparities in Testing | Baseline through study completion (26 months)
  Explore impact on testing disparities by race/ethnicity and SES

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Belinda E Reininger, DrPh, Principal Investigator — The University of Texas Health Science Center, Brownsville; David D McPherson, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Paul McGaha, DO, Principal Investigator — The University of Texas Health Science Center, Tyler; Marcia C de Oliveira Otto, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Kayo Fujimoto, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - The University of Texas Health Science Center, Brownsville, Brownsville, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No